CLINICAL TRIAL: NCT04153539
Title: Acute Health Effects of Traffic-Related Air Pollution Exposure Among Healthy Young Adults: A Randomized, Crossover Trial
Brief Title: Acute Health Effects of Traffic-Related Air Pollution Exposure
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haidong Kan, Professor, Fudan University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: FDUEH-6
Record Dates: First submitted 2019-11-03; First posted 2019-11-06 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Cardiovascular System; Respiratory System
Keywords: Traffic-related pollution; Randomized controlled trial; Acute health effects
MeSH Terms: interventions — Walking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walking along a busy road (Experimental): Participants in this group will be asked to walk along a busy road for 4.5 hours.
  Interventions: Behavioral: Walking along a busy road
- Walking in a traffic-free park (Active Comparator): Participants in this group will be asked to walk in a traffic-free park for 4.5 hours.
  Interventions: Behavioral: Walking in a traffic-free park

INTERVENTIONS:
Behavioral: Walking along a busy road — The intervention group will walk along a busy road and be exposed to traffic-related air pollution for 4.5 hours (from 13:00 to 17:30), while alternating 15-minute walking and 30-minute rest periods.
  Arms: Walking along a busy road
Behavioral: Walking in a traffic-free park — The control group will walk in a traffic-free park for 4.5 hours (from 13:00 to 17:30), while alternating 15-minute walking and 30-minute rest periods.
  Arms: Walking in a traffic-free park

SUMMARY:
This study aims to assess the effects of acute exposure to traffic-related air pollution and the underlying mechanisms.

DETAILED DESCRIPTION:
The investigators will conduct a randomized, crossover trial among 72 healthy young adults in Shanghai, China. The eligible participants will be randomly divided into 2 groups (36 volunteers per group). During the first stage, participants will be requested to take one walking task (from 13:00 to 17:30). The exposed group will walk along a busy road and be exposed to traffic-related air pollution, while the control group will walk in a traffic-free park. During the first 3 hours, all participants will rest for 30 minutes after each 15-minute walking. From 16:00, participants will stop walking and rest for 1.5 hours. Then both groups will enter a 2-week washout period. In the second stage, there will also be one walking task (from 13:00 to 17:30). The two groups will exchange their walking sites and repeat the previous trial. Physical examinations will be performed both before and after each walking task. Besides, we will ask volunteers to stay in school during the two days before walking. Health examinations include symptoms questionnaires, blood pressure tests, Holter monitoring, and spirometry. We plan to collect blood, urine, oropharyngeal swabs, and exhaled breath condensate before exposure, about one hour after exposure, and next morning.

ELIGIBILITY:
Inclusion Criteria:

* Living in Shanghai during the study period;
* Body mass index > 18.5 and ≤ 28;
* Non-smoking, no history of alcohol or drug abuse;
* Completing the walking task we required.

Exclusion Criteria:

* Current or ever smokers;
* Subjects with allergic disease, such as allergic rhinitis, allergic asthma, and atopy;
* Subjects with cardiovascular disease, such as congenital heart disease, pulmonary heart disease, and hypertension;
* Subjects with respiratory disease, such as asthma, chronic bronchitis, and chronic obstructive pulmonary disease;
* Subjects wih chronic disease, such as diabetes, chronic hepatitis, and kidney disease;
* Subjects with a history of major surgery;
* Abnormal spirometry (FEV1 and FVC ≤ 75% of predicted and FEV1/FVC ≤ 0.65);
* Medication use or dietary supplements intake in recent two months;

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2019-12-08 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in FEV1 | FEV1 will be examined before exposure, half an hour after exposure and 12 hours after exposure.
  We plan to measure changes in forced expiratory volume in 1 second.
Blood Pressure | Blood pressure will be measured for 24 hours from 8:00 am on the morning of intervention to 8:00 am on the next morning.
  We plan to measure systolic blood pressure (SBP) and diastolic blood pressure (DBP).
Heart Rate Variability Parameters | Volunteers will be asked to wear electrographic Holter monitors for 24 hours from 8:00 am on the morning of intervention to 8:00 am on the next morning.
  We plan to measure heart rate variability (HRV) parameters.

SECONDARY OUTCOMES:
Changes of FVC | 7:00 AM on the day of the walking session, half an hour after exposure and 12 hours after exposure (next morning)
  Changes of forced vital capacity
Changes of FEV1/FVC | 7:00 AM on the day of the walking session, half an hour after exposure and 12 hours after exposure (next morning)
  Changes of the ratio of forced expired volume in 1 second (FEV1) to forced vital capacity (FVC)
Changes of MMEF | 7:00 AM on the day of the walking session, half an hour after exposure and 12 hours after exposure (next morning)
  Changes of maximal mid-expiratory flow

OTHER OUTCOMES:
Differences in DNA methylation levels detected in whole-blood between the two exposures | 1 hour after the end of the exposure session
  Genome-wide DNA methylation in whole-blood were detected using Illumina 850K Beadchip. The study is to identify differential CpG loci after TRAP exposure
Differences in exosome RNA expression levels detected in plasma transcriptomics between the two exposures | 1 hour after the end of the exposure session
  Illumina-based transcriptomics is non-targeted. The study is to find the differentially expressed exosome RNA in plasma after TRAP exposure
Differences in exosome miRNA expression levels detected in plasma transcriptomics between the two exposures | 1 hour after the end of the exposure session
  Illumina-based transcriptomics is non-targeted. The study is to find the differentially expressed exosome miRNA in plasma after TRAP exposure
Differences in protein levels detected in plasma proteomics between the two exposures | 1 hour after the end of the exposure session
  Mass spectrometry-based plasma proteomics is non-targeted. The study is to find the differentially expressed proteins in plasma after TRAP exposure
Differences in metabolic profiling detected in serum mass spectrometry-based non-targeted metabolomics between the two exposures | 1 hour after the end of the exposure session
  The study is to explore the differential metabolic profiling in serum after TRAP exposure.
Differences in metabolic profiling detected in urine mass spectrometry-based non-targeted metabolomics between the two exposures | 1 hour after the end of the exposure session
  The study is to explore the differential metabolic profiling in urine after TRAP exposure.
Differences in lipids levels detected in serum lipidomics between the two exposures | 1 hour after the end of the exposure session
  Mass spectrometry-based serum lipids is non-targeted. The study is to find the differential lipids in serum between the road scenario and the park scenario
Differences in protein levels detected in targeted serum proteomic chip between the two exposures | 1 hour after the end of the exposure session
  Targeted serum proteomic chip was conducted using the RayBio Biotin Label-based Human Antibody Array, which covers a total of 507 human proteins, including cytokines, inflammatory proteins, growth factors, cell adhesion molecules, soluble receptors and chemokines, and proteins related to angiogenesis and atherosclerosis. The study is to find the differential proteins in serum between the road scenario and the park scenario
Differences in metabolic profiling detected in airway mass spectrometry-based non-targeted metabolomics between the two exposures | 1 hour after the end of the exposure session
  The study is to explore the differential metabolic profiling in exhaled breath condensate after TRAP exposure.
Change in CRP concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session, and 7:00 AM in the next morning
  Change in the serum concentrations of C-reactive protein
Change in ITAC concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session, and 7:00 AM in the next morning
  Change in the serum concentrations of Interferon-induced T-cell alpha chemoattractant
Change in GM-CSF concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session, and 7:00 AM in the next morning
  Change in the serum concentrations of Granulocyte-macrophage colony-stimulating factor
Change in IFN-gamma concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session, and 7:00 AM in the next morning
  Change in the serum concentrations of Interferon-gamma
Change in IL-10 concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session, and 7:00 AM in the next morning
  Change in the serum concentrations of Interlukin-10
Change in IL-17A concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session, and 7:00 AM in the next morning
  Change in the serum concentrations of Interleukin-17A
Change in IL-1 beta concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session, and 7:00 AM in the next morning
  Change in the serum concentrations of Interlukin-1 beta
Change in IL-23 concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session, and 7:00 AM in the next morning
  Change in the serum concentrations of Interleukin-23
Change in IL-6 concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session, and 7:00 AM in the next morning
  Change in the serum concentrations of Interleukin-6
Change in IL-8 concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session, and 7:00 AM in the next morning
  Change in the serum concentrations of Interleukin-8
Change in TNF alpha concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session, and 7:00 AM in the next morning
  Change in the serum concentrations of Tumor necrosis factor-α
Change in MDA concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session, and 7:00 AM in the next morning
  Change in the serum concentrations of Malondialdehyde
Change in 8-OH-DG concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session, and 7:00 AM in the next morning
  Change in the urine concentrations of 8-hydroxy-2'-deoxyguanosine
Change in ACE concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session
  Change in the serum concentrations of Angiotensin converting enzymes
Change in Angiotensin II concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session
  Change in the serum concentrations of Angiotensin II
Change in ALD concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session
  Change in the urine concentrations of Aldosterone
Change in TF concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session
  Change in the serum concentrations of Tissue factor
Change in Fibrinogen concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session
  Change in the serum concentrations of Fibrinogen
Change in PAI-1 concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session
  Change in the serum concentrations of Plasminogen Activator inhibitor-1
Change in vWF concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session
  Change in the serum concentrations of von Willebrand factor
Change in CRF concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session, and 7:00 AM in the next morning
  Change in the serum concentrations of Corticotropin-Releasing Factor
Change in ACTH concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session, and 7:00 AM in the next morning
  Change in the serum concentrations of Adrenocorticotropic hormone
Change in Cortisol concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session, and 7:00 AM in the next morning
  Change in the serum concentrations of Cortisol
Change in Cholesterol concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session, and 7:00 AM in the next morning
  Change in the serum concentrations of Cholesterol
Change in TAG concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session, and 7:00 AM in the next morning
  Change in the serum concentrations of Triglyceride
Change in LDL-C concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session, and 7:00 AM in the next morning
  Change in the serum concentrations of Low-density lipoprotein cholesterol
Change in Glucose concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session, and 7:00 AM in the next morning
  Change in the serum concentrations of Glucose
Change in Insulin concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session, and 7:00 AM in the next morning
  Change in the serum concentrations of Insulin
Changes in SP-D concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session
  Change in the serum concentrations of surfactant proteins D
Changes in Ezrin concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session
  Change in the exhaled breath condensate concentrations of Ezrin
Changes in 8-isoprostane concentrations between the two exposures | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session
  Change in the exhaled breath condensate concentrations of 8-isoprostane
Changes in TNF-α concentrations | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session
  Change in the exhaled breath condensate concentrations of tumor necrosis factor-α
Changes of the scores of respiratory symptoms questionnaires | 7:00 AM on the day of the walking session, 1 hour after the end of the exposure session
  Changes of scores of respiratory symptoms questionnaires both the total and each symptom specified

CONTACTS AND LOCATIONS:
Overall Officials: Haidong Kan, PhD, Study Director — Department of Environmental Health, School of Public Health, Fudan University
Locations (1):
- Department of Environmental Health, School of Public Health, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No